CLINICAL TRIAL: NCT05439798
Title: Comparison of the Effects of Palonosetron + Dexamethazone, Ondansetron + Dexamethazone and Dexametazone Alone Against Postoperative Nausea and Vomiting in Pediatric Patients Undergoing Laparoscopic Surgery
Brief Title: Effect of Palonosetron, Ondansetron and Dexamethasone in the Prevention of Postoperative Nausea and Vomiting
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Faruk Cicekci, Associate Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: farukcicekci6
Record Dates: First submitted 2022-05-18; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Laparoscopic Surgery; Pediatrics; Nausea and Vomiting, Postoperative; Antiemetics; Therapeutic Use
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blind, controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group OD (Group ondansetron+dexamethasone) (Active Comparator): The patients in Group OD (Group ondansetron+dexamethasone) will be given intravenous (iv) ondansetron (0.1 mg.kg-1) + dexamethasone (0.5 mg.kg-1).
  Interventions: Drug: Ondansetron+Dexamethasone
- Group PD (Group palonosetron+dexamethasone) (Active Comparator): The patients in Group PD (Group palonosetron+dexamethasone) will be given intravenous (iv) palonosetron (0.75µg.kg-1) + dexamethasone (0.5 mg.kg-1).
  Interventions: Drug: Palonosetron+Dexamethasone
- Group D (Group Dexamethasone) (Placebo Comparator): The patients in Group D (Group Dexamethasone) will be given intravenous (iv) dexamethasone (0.5 mg.kg-1).
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Ondansetron+Dexamethasone — The patients in Group OD (Group ondansetron+dexamethasone) will be given intravenous (iv) ondansetron (0.1 mg.kg-1) + dexamethasone (0.5 mg.kg) The patients in Group PD (Group palonosetron+dexamethasone) will be given intravenous (iv) palonosetron (0.75µg.kg-1) + dexamethasone (0.5 mg.kg-1).
  The patients In Group D (Group Dexamethasone) will be given iv only dexamethasone (0.5 mg.kg-1)
  Arms: Group OD (Group ondansetron+dexamethasone)
Drug: Palonosetron+Dexamethasone — The patients in Group OD (Group ondansetron+dexamethasone) will be given intravenous (iv) ondansetron (0.1 mg.kg-1) + dexamethasone (0.5 mg.kg) The patients in Group PD (Group palonosetron+dexamethasone) will be given intravenous (iv) palonosetron (0.75µg.kg-1) + dexamethasone (0.5 mg.kg-1).
  The patients In Group D (Group Dexamethasone) will be given iv only dexamethasone (0.5 mg.kg-1)
  Arms: Group PD (Group palonosetron+dexamethasone)
Drug: Dexamethasone — Dexamethasone
  Arms: Group D (Group Dexamethasone)

SUMMARY:
Postoperative nausea and vomiting (PONV) is an important outcome for the patient; patients generally rate PONV as worse than postoperative pain. The term PONV is typically used to describe nausea and/or vomiting or retching in the post-anesthetic care unit or within 24 hours postoperatively. Postoperative nausea and vomiting usually resolves or is treated without sequelae, but may require unexpected hospitalization and delay recovery room discharge. In the prophylaxis of PONV, ondansetron is one of the first widely used 5-HT3 receptor antagonists. Palonosetron, on the other hand, is a second generation 5-HT3 receptor antagonist with a half-life of 40 hours and higher receptor binding affinity. In addition, dexamethasone is another class of drugs that has emerged as a potentially useful prophylaxis for patients who are a corticosteroid and are at high risk of PONV with minimal side effects. However, a multimodal approach rather than antiemetic prophylaxis with a single pharmacological agent is described as a good way to reduce PONV, especially in high-risk cases. Conducted a previous systematic review and meta-analysis of the addition of dexamethasone to various 5-HT3 antagonists; however, it included only one study of palonosetron + dexamethasone. Since then, several meta-analyses have been performed on the efficacy of the combination of palonosetron and dexamethasone. This study was designed to find out the incidence of PONV by comparing the efficacy of the combination of palonosetron-dexamethasone, ondansetron-dexamethasone and dexamethasone alone for the prevention of PONV in patients undergoing pediatric laparoscopic surgery.

DETAILED DESCRIPTION:
This study will be conducted with the data to be obtained from the Anesthesiology Surgery Form and Pediatric Surgery Service Forms in 66 patients aged 7-18 years, after the approval of Local Ethics Committee, Faculty of Medicine, Selcuk University. The patıents will be randomized ınto 3 groups. Patients in Group OD (n = 22) (Group ondansetron+dexamethasone) will be given intravenous (iv) ondansetron (0.1 mg.kg-1) + dexamethasone (0.5 mg.kg-1). For this group of patients, ondansetron (0.1 mg.kg-1) (5 ml) will be prepared and will be named No: 1. It will be administered at the 8th and 16th hours postoperatively. In Group PD (n = 22) (Group palonosetron+dexamethasone), patients will be given intravenous (iv) palonosetron (0.75µg.kg-1) + dexamethasone (0.5 mg.kg-1). In Group D (n = 22) (Group Dexamethasone) iv only dexamethasone (0.5 mg.kg-1) will be given. For the patients in Group PD and Group D, normal saline (SF) (5 ml solution) will be prepared for intravenous administration and will be named No: 2 and 3, respectively, and will be administered again at the 8th and 16th hours. The reason why we give SF here is to provide drug blanking, but not to give active drug, since the half-life of palonasetron and dexamethasone is long, up to 36 hours. The files of the patients will be examined and demographic data. For the primary purpose of this study, PONV values will be evaluated at 2, 6, 12, 24, 48, and 72 hours postoperatively. The intensity of nausea (0 = no nausea, 10 = worst possible nausea) will be rated on a verbal numerical rating scale (VNRS). The severity of nausea and vomiting will be classified as mild (1-3), moderate (4-6) and severe (7-10) according to VNRS scores. Secondary endpoints, time of taking first rescue antiemetic and total dose of rescue antiemetic, and complications (dizziness, headache, and arrhythmia) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class I-II,
* Between the ages of 7-18,
* Patients with written informed consent from themselves and their parents

Exclusion Criteria:

* Allergic to study drugs,
* Taking antiemetic drugs 24 hours before the operation,
* Gastroesophageal reflux disease,
* Body mass index (BMI) >35 kg/m 2,
* In the period of menstruation,
* Receiving cancer chemotherapy in the last four weeks,
* Allergy to NSAIDs,
* Patients with bronchial asthma

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of palonosetron, ondansetron and dexamethasone in postoperative nausea and vomiting | 72 hours
  The primary endpoint of this study was to find the incidence of PONV among the three groups.

SECONDARY OUTCOMES:
The time to first rescue antiemetic intake | 72 hours
  The Secondary endpoints were the time to first rescue antiemetic intake
The total amount of antiemetic use | 72 hours
  the total amount of antiemetic use
The complications | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)